CLINICAL TRIAL: NCT07127718
Title: Decreasing Leptospirosis Emergence Through Prognosis and Treatment Optimization (DeLEPTO) Project 1: Preventive Strategies for Early and Late Complications of Leptospirosis
Brief Title: Preventive Strategies for Early and Late Complications of Leptospirosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Kidney and Transplant Institute, Philippines (Other)
Collaborators: San Lazaro Hospital, Philippines (Unknown); Institute of Human Genetics, National Institutes of Health - University of the Philippines Manila, Philippines (Unknown); Department of Science and Technology, Philippines (Unknown)
Responsible Party: Principal Investigator, Romina A. Danguilan, Deputy Executive Director for Medical Services, National Kidney and Transplant Institute, Philippines
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJREB 2024-70
Record Dates: First submitted 2025-07-16; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Leptospirosis
Keywords: leptospirosis; plasma transfusion; hemoperfusion; extracorporeal membrane oxygenation; complement factor I; CFI; complications; renal complications; pulmonary complications
MeSH Terms: conditions — Leptospirosis | interventions — Hemoperfusion; Extracorporeal Membrane Oxygenation; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Prophylactic Plasma Component Therapy with Conventional Treatment (PPTTRT) (Experimental): This serves as the case arm for prophylactic plasma transfusion (PPT).
  Participants in the PPTTRT arm will receive transfusion if the peripheral blood mononuclear cell (PBMC) complement factor I (CFI) quantitative real-time polymerase chain reaction (qPCR) deltaCT is found to be at least 25 or more. These participants will also be receiving standard of care treatment.
  Participants in the PPTTRT arm with PBMC CFI qPCR deltaCT less than 25 will only be receiving standard of care treatment.
  If a participant is found to have a Murray score of greater than or equal to 2.75 over the course of the hospital stay, they will undergo extracorporeal membrane oxygenation (ECMO).
  Interventions: Biological: Prophylactic Plasma Transfusion; Device: Extracorporeal Membrane Oxygenation; Other: Conventional therapy
- Conventional Treatment (PPTCONV) (Active Comparator): This serves as the control arm for prophylactic plasma transfusion (PPT).
  Participants in the PPTCONV arm will only be receiving standard of care treatment.
  If a participant is found to have a Murray score of greater than or equal to 2.75 over the course of the hospital stay, they will undergo extracorporeal membrane oxygenation (ECMO).
  Interventions: Device: Extracorporeal Membrane Oxygenation; Other: Conventional therapy
- Hemoperfusion Treatment with Conventional Treatment (HPTRT) (Experimental): This serves as the case arm for hemoperfusion (HP).
  Participants in the HPTRT arm will receive hemoperfusion and standard of care.
  Participants with a Murray score of greater than or equal to 2.75 will undergo extracorporeal membrane oxygenation (ECMO) as a rescue treatment.
  Interventions: Device: Hemoperfusion; Device: Extracorporeal Membrane Oxygenation; Other: Conventional therapy
- Conventional Treatment (HPCONV) (Active Comparator): This serves as the control arm for hemoperfusion (HP).
  Participants in the HPCONV arm will only be receiving standard of care.
  Participants with a Murray score of greater than or equal to 2.75 will undergo extracorporeal membrane oxygenation (ECMO) as a rescue treatment.
  Interventions: Device: Extracorporeal Membrane Oxygenation; Other: Conventional therapy

INTERVENTIONS:
Biological: Prophylactic Plasma Transfusion — ABO/Rh-type compatible fresh frozen plasma (FPP) units will be thawed to 37° prior to administration. Plasma transfusion will be administered intravenously, 1 unit for 4 hours every 12 hours. There will be two consecutive days for the transfusion for a total of 4 units.
  Other Names: Prophylactic Plasma Component Transfusion; Plasma Transfusion; Prophylactic Plasma Component Therapy; PPT
  Arms: Prophylactic Plasma Component Therapy with Conventional Treatment (PPTTRT)
Device: Hemoperfusion — The hemoperfusion (HP) procedure will follow the standard procedure of National Kidney and Transplant Institute (NKTI) using Jafron HA330 hemoperfusion cartridge. First, an internal jugular catheter is attached to the patient. Alternatively, an arteriovenous fistula or arteriovenous graft may be placed on the patient. The patient will then be hooked to a hemodialysis machine. Blood pump speed will be set to 150-200mL/min, and HP will last for 2 to 2.5 hours. Whole blood will flow through the sorbent HA330 cartridge and back to the patient. Anticoagulation is not necessary due to the short treatment time. Hemoperfusion will be repeated after 12-24 hours for at least three days.
  Other Names: HP
  Arms: Hemoperfusion Treatment with Conventional Treatment (HPTRT)
Device: Extracorporeal Membrane Oxygenation — A veno-venous ECMO (VV ECMO) will be applied by aseptically inserting a venous cannula into the femoral veins. The patients will be hooked to an ECMO machine. Patients without significant bleeding or vascular intervention will be managed with an activated clotting time set at 140-180 sec by 800-1000 U/h of heparin. Otherwise, heparin will be titrated to maintain a partial thromboplastin time of 60-80 sec.
  ECMO settings are as follows:
  * Mean blood pressure of >60 mm
  * SaO2 at >90% with a flow of 3.5-4.5 L/min
  * Hematocrit at >35%
  * Platelets >50000-100000/mL
  * Transfusions will be done when necessary
  Criteria for weaning:
  * ABG:
    * pH 7.35-7.45
    * PaO2 >80 mm Hg
    * PCO2 <45 mm Hg
  * Under the following conditions:
    * Gas blender FiO2 of 0.21
    * Sweep gas of 0 L/min at an ECMO flow of 2 L/min
    * Ventilator mode (if applicable):
      * FiO2 of 0.6
      * Tidal volume of 6 mL/kg
      * PEEP of 8 cmH2O
      * RR of 12-16/min for VV ECMO or 3 L/min of O2 via nasal prong with awakening ECMO patients
  Other Names: ECMO
Other: Conventional therapy — Conventional therapy for leptospirosis includes antibiotics, fluids, inotropes, renal replacement therapy, ventilator support, and other treatment that the attending physician deems necessary.
  Other Names: Standard of care

SUMMARY:
The goal of this clinical trial is to learn if complement factor I (CFI) works to predict development of complications in participants with leptospirosis. It will also learn if plasma transfusion, hemoperfusion, and extracorporeal membrane oxygenation works to treat participants with leptospirosis. The main questions it aims to answer are:

* Does a low level of CFI predict the development of lung damage in participants with leptospirosis?
* Does plasma tranfusion lower the chances of participants getting lung damage from leptospirosis?
* Does hemoperfusion work to remove harmful materials from the blood of participants with leptospirosis?
* Does extracorporeal membrane oxygenation increase the chance of survival in participants with lung damage?

Researchers will compare plasma tranfusion and hemoperfusion to conventional therapy (standard of care for leptospirosis, including antibiotics, fluids, and other treatment that the doctor deems necessary) to see if these novel therapies work to treat leptospirosis.

Participants will:

* Give blood samples for the study of CFI
* Receive conventional therapy and/or plasma transfusion for 4 times in 2 days, OR
* Receive conventional therapy and/or hemoperfusion for at least 3 days, AND/OR
* Receive extracorporeal membrane oxygenation if their condition worsens

DETAILED DESCRIPTION:
This study aims to determine the clinical utility of complement factor I (CFI) as a prognosticator in patients with complicated leptospirosis without severe pulmonary complications and to determine if its guidance to preemptive measures can lead to a reduction in adverse clinical outcomes, specifically the occurrence of pulmonary bleeding and acute respiratory distress syndrome (ARDS), and mortality. Hence, the results of the study may lead to novel treatment approaches that can be readily applied in clinical practice. The decision to provide preemptive non-invasive therapies or early intensive care admission could lead to significant breakthroughs in managing the disease.

Within the Decreasing Leptospirosis Emergence through Prognosis and Treatment Optimization (DeLEPTO) program's vision of developing tools to increase the survival of leptospirosis patients, this project will explore the avenue of novel tertiary care. Specifically, the program will look into the possibility of CFI repletion using plasma transfusion, cytokine depletion strategies using hemoperfusion (HP), and extracorporeal membrane oxygenation (ECMO). It would be interesting to see how such interventions could work individually or in a pipeline with other proposed interventions. In addition to plasma therapy, ECMO was observed to improve outcomes in severe leptospirosis. As a secondary endpoint, it would also be interesting to know if CFI can prognosticate who will benefit the most from such interventions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with acute fever (38ºC for at least two days) and at least one of the following: myalgia, jaundice, headache, meningeal irritation, oliguria, conjunctival suffusion
* Who have a microscopic agglutination test (MAT) that indicates a single serum sample MAT titer greater than or equal to 1:400
* Or a positive result for the latex agglutination test or a repeat test after seven days
* Or a positive blood culture of leptospira WITHOUT the complication specified in a subgroup of interest
* PPTTRT/PPTCONV: Not requiring ventilator support
* HPTRT/HPCONV: Dialysis Requiring Acute Kidney Injury. Defined as KDIGO Acute Kidney Injury Stage 3 or requiring renal replacement therapy to correct intractable acidosis, electrolyte abnormality, or over uremic encephalopathy or pericarditis
* HPTRT/HPCONV: Vasopressor Requiring - The subject must have received intravenous fluid resuscitation of a minimum of 30ml/kg within 24 hours of eligibility and still with hypotension (blood pressure less than 90/60, MAP less than 65) requiring vasopressor support
* HPTRT/HPCONV: SOFA SCORE less than 15
* ECMO: A Murray score of greater than or equal to 2.75

Exclusion Criteria:

* Previous diagnosis of chronic kidney disease or on maintenance dialysis
* Previous diagnoses of diseases associated with hemoptysis, such as bronchiectasis
* Blood dyscrasias, malignancy, severe heart disease, HIV, cavitary PTB, Cirrhosis by ultrasound, severe malnutrition (Weight of less than 35kg)
* Post cardiac arrest or those with GCS <8 at present. Participant has had chest compressions or CPR
* Pregnancy
* PPTTRT/PPTCONV: Requiring emergent dialyses
* PPTTRT/PPTCONV: Significant renal impairment as defined by eGFR less than 30
* PPTTRT/PPTCONV: Significant lung pathology as defined by P/F ratio less than 300, or obvious respiratory distress
* PPTTRT/PPTCONV: Presence of severe neurological symptoms
* PPTTRT/PPTCONV: Hypotension (or need for vasopressor support)
* PPTTRT/PPTCONV: Ongoing hemodynamic instability

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 678 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Determination of CFI levels via qPCR and via ELISA | At baseline and Day 1 post-treatment, assessed up to study completion, an average of 3 years
  Baseline blood samples will be obtained for CFI qPCR and ELISA upon enrollment. Post-treatment blood samples will be obtained for ELISA. Correlation of values of qPCR results to ELISA data will be performed using Pearson correlation (r2 of 0.80 or higher will be considered highly correlated). Test for concordance using Kendall's W will be done.
Hospital Days | From admission to discharge from the hospital, assessed up to study completion, an average of 3 years
  Hospital days will be computed from the date of admission to the date of discharge. Mortality or discharge against medical advice will be penalized with a maximum stay of at least 30 days.
Occurrence of Mortality | From admission to discharge from the hospital or date of death, assessed up to study completion, an average of 3 years
  Mortality is defined as death occurring to be related to the natural course of the present condition of leptospirosis or its complication, but not more than two weeks upon discharge by attending physician after being assessed as well recovered, or the like.
Presence of Significant Pulmonary Involvement | From admission to discharge from the hospital, assessed up to study completion, an average of 3 years
  As in leptospirosis (Weil's syndrome) plus evidence of pulmonary injury as indicated by (1) the need for mechanical ventilator support, (2) P/F ratio <200,(3) gross hemoptysis, OR (4) chest x-ray result consistent with leptospirosis-related pulmonary changes.

SECONDARY OUTCOMES:
Need for Renal Replacement Therapy | From admission to discharge from the hospital, assessed up to study completion, an average of 3 years
  Number of days requiring dialysis during hospital stay.
Need for Inotropic Support | From admission to discharge from the hospital, assessed up to study completion, an average of 3 years
  Number of days requiring inotropic support to attain MAP >65 and number of days requiring each inotrope
Need for Emergent Invasive Respiratory Support | From admission to discharge from the hospital, assessed up to study completion, an average of 3 years
  Inability to maintain Sp02 >92% on maximum non-invasive respiratory support
Presence of Refractory Hypotension | From admission to discharge from the hospital, assessed up to study completion, an average of 3 years
  Occurrence of systolic blood pressure less than 90 mm Hg, OR mean arterial pressure less than 65 mm Hg, OR a decrease of 40 mm Hg in systolic blood pressure compared to baseline: unresponsive to crystalloid ﬂuid challenge of 20 to 40 mL/kg OR requiring vasopressor support
Presence of Significant Renal Involvement | From admission to discharge from the hospital, assessed up to study completion, an average of 3 years
  As in leptospirosis (Weil's syndrome), plus evidence of severe acute kidney injury as indicated by the need for emergency dialysis due to intractable acidosis, hyperkalemia, uremic encephalopathy or pericarditis.
Need for Extracorporeal Membrane Oxygenation (ECMO) assessed via Murray score | From admission to discharge from the hospital, assessed up to study completion, an average of 3 years
  A participant is considered for Extracorporeal Membrane Oxygenation (ECMO) when he/she attains a Murray score of greater than or equal to 2.75.
  The Murray score is a scale used to assess the severity of acute lung injury in acute respiratory distress syndrome (ARDS). A Murray score of 0 means there is no lung injury; a score of 0.1-2.5 means there is mild to moderate lung injury; and a score of greater than 2.5 means there is severe lung injury.
Need for Extracorporeal Membrane Oxygenation (ECMO) assessed via Horowitz Index for Lung Function (P/F Ratio) | From admission to discharge from the hospital, assessed up to study completion, an average of 3 years
  A participant is considered for Extracorporeal Membrane Oxygenation (ECMO) when he/she attains the a Horowitz Index for Lung Function (P/F Ratio) of less than 200.
  The Horowitz Index for Lung Function (P/F Ratio) is the ratio of arterial oxygen partial pressure (PaO2) and the fractional inspired oxygen (FiO2). A P/F ratio of greater than 300 mmHg indicates absence of ARDS; 201-300 mmHg is mild ARDS; 101-200 mmHg is moderate ARDS; and less than or equal to 100 is severe ARDS.
Intensive Care Unit (ICU) Days | From admission into ICU to date out of ICU, assessed up to study completion, an average of 3 years
  Number of days patient is required to stay in ICU (date out of ICU will be date ordered by the attending physician)

CONTACTS AND LOCATIONS:
Overall Officials: Romina A Danguilan, MD, Principal Investigator — National Kidney and Transplant Institute, Philippines
Locations (3):
- Philippines (3):
  - Institute of Human Genetics, National Institutes of Health - University of the Philippines Manila, Manila, National Capital Region
  - San Lazaro Hospital, Manila, National Capital Region
  - National Kidney and Transplant Institute, Quezon City, National Capital Region

IPD SHARING:
Plan to Share IPD: Yes
The patient information will not be shared at present as the study is still ongoing and there is intellectual property involved. However, general IPD, such as age, sex, and affliction, will be shared, together with important clinical outcomes such as mortality and incidence of renal and or pulmonary complications, only after appropriate intellectual property protection.

REFERENCES:
- [Background] Milhem MM, Knutson T, Yang S, Zhu D, Wang X, Leslie KK, Meng X. Correlation of MTDH/AEG-1 and HOTAIR Expression with Metastasis and Response to Treatment in Sarcoma Patients. J Cancer Sci Ther. 2011 Dec 29;S5(4):004. PMID 23543869
- [Background] Popugaev KA, Bakharev SA, Kiselev KV, Samoylov AS, Kruglykov NM, Abudeev SA, Zhuravel SV, Shabanov AK, Mueller T, Mayer SA, Petrikov SS. Clinical and pathophysiologic aspects of ECMO-associated hemorrhagic complications. PLoS One. 2020 Oct 13;15(10):e0240117. doi: 10.1371/journal.pone.0240117. eCollection 2020. PMID 33048966
- [Background] Na SJ, Chung CR, Choi HJ, Cho YH, Sung K, Yang JH, Suh GY, Jeon K. The effect of multidisciplinary extracorporeal membrane oxygenation team on clinical outcomes in patients with severe acute respiratory failure. Ann Intensive Care. 2018 Feb 27;8(1):31. doi: 10.1186/s13613-018-0375-9. PMID 29484504
- [Background] Combes A, Brodie D, Bartlett R, Brochard L, Brower R, Conrad S, De Backer D, Fan E, Ferguson N, Fortenberry J, Fraser J, Gattinoni L, Lynch W, MacLaren G, Mercat A, Mueller T, Ogino M, Peek G, Pellegrino V, Pesenti A, Ranieri M, Slutsky A, Vuylsteke A; International ECMO Network (ECMONet). Position paper for the organization of extracorporeal membrane oxygenation programs for acute respiratory failure in adult patients. Am J Respir Crit Care Med. 2014 Sep 1;190(5):488-96. doi: 10.1164/rccm.201404-0630CP. PMID 25062496
- [Background] Cheng R, Hachamovitch R, Kittleson M, Patel J, Arabia F, Moriguchi J, Esmailian F, Azarbal B. Complications of extracorporeal membrane oxygenation for treatment of cardiogenic shock and cardiac arrest: a meta-analysis of 1,866 adult patients. Ann Thorac Surg. 2014 Feb;97(2):610-6. doi: 10.1016/j.athoracsur.2013.09.008. Epub 2013 Nov 8. PMID 24210621
- [Background] Khalid N, Javed H, Ahmad SA, Edelman JJ, Shlofmitz E, Chen Y, Musallam A, Rogers T, Hashim H, Bernardo NL, Waksman R. Analysis of the Food and Drug Administration Manufacturer and User Facility Device Experience Database for Patient- and Circuit-Related Adverse Events Involving Extracorporeal Membrane Oxygenation. Cardiovasc Revasc Med. 2020 Feb;21(2):230-234. doi: 10.1016/j.carrev.2019.11.011. Epub 2019 Nov 20. PMID 31767523
- [Background] Xu L, Wu X, Zou Y. Clinical efficacy comparison of HA280 and DNA280 immunoadsorption column in treating systemic lupus erythematosus. Mod Rheumatol. 2016;26(1):94-8. doi: 10.3109/14397595.2015.1056955. Epub 2015 Aug 19. PMID 26025438
- [Background] Pomare Montin D, Ankawi G, Lorenzin A, Neri M, Caprara C, Ronco C. Biocompatibility and Cytotoxic Evaluation of New Sorbent Cartridges for Blood Hemoperfusion. Blood Purif. 2018;46(3):187-195. doi: 10.1159/000489921. Epub 2018 Jun 8. PMID 29886501
- [Background] Semple JW, Rebetz J, Kapur R. Transfusion-associated circulatory overload and transfusion-related acute lung injury. Blood. 2019 Apr 25;133(17):1840-1853. doi: 10.1182/blood-2018-10-860809. Epub 2019 Feb 26. PMID 30808638
- [Background] Vlaar AP, Juffermans NP. Transfusion-related acute lung injury: a clinical review. Lancet. 2013 Sep 14;382(9896):984-94. doi: 10.1016/S0140-6736(12)62197-7. Epub 2013 May 1. PMID 23642914
- [Background] Popovsky MA. Transfusion-associated circulatory overload: the plot thickens. Transfusion. 2009 Jan;49(1):2-4. doi: 10.1111/j.1537-2995.2008.02010.x. No abstract available. PMID 19140808
- [Background] Chowdary P, Saayman AG, Paulus U, Findlay GP, Collins PW. Efficacy of standard dose and 30 ml/kg fresh frozen plasma in correcting laboratory parameters of haemostasis in critically ill patients. Br J Haematol. 2004 Apr;125(1):69-73. doi: 10.1111/j.1365-2141.2004.04868.x. PMID 15015971
- [Background] Alam A, Lin Y, Lima A, Hansen M, Callum JL. The prevention of transfusion-associated circulatory overload. Transfus Med Rev. 2013 Apr;27(2):105-12. doi: 10.1016/j.tmrv.2013.02.001. Epub 2013 Mar 1. PMID 23465703
- [Background] Arokianathan D, Trower K, Pooboni S, Sosnowski A, Moss P, Thaker H. Leptospirosis: a case report of a patient with pulmonary haemorrhage successfully managed with extra corporeal membrane oxygenation. J Infect. 2005 Feb;50(2):158-62. doi: 10.1016/j.jinf.2004.09.010. PMID 15667919
- [Background] Kahn JM, Muller HM, Kulier A, Keusch-Preininger A, Tscheliessnigg KH. Veno-arterial extracorporeal membrane oxygenation in acute respiratory distress syndrome caused by leptospire sepsis. Anesth Analg. 2006 May;102(5):1597-8. doi: 10.1213/01.ANE.0000215121.67833.2F. No abstract available. PMID 16632865
- [Background] Liao CY, Ben RJ, Wu HM, Chang SK, Liu MY, Chin HK, Yeh YC. Acute Respiratory Distress Syndrome Manifested by Leptospirosis Successfully Teated by Extracorporeal Membrane Oxygenation (ECMO). Intern Med. 2015;54(22):2943-6. doi: 10.2169/internalmedicine.54.4528. Epub 2015 Nov 15. PMID 26568015
- [Background] Pardinas M, Mendirichaga R, Budhrani G, Garg R, Rosario L, Rico R, Panos A, Baier H, Krick S. Use of Aminocaproic Acid in Combination With Extracorporeal Membrane Oxygenation in a Case of Leptospirosis Pulmonary Hemorrhage Syndrome. Clin Med Insights Circ Respir Pulm Med. 2017 Mar 2;11:1179548416686068. doi: 10.1177/1179548416686068. eCollection 2017. PMID 28469503
- [Background] Umei N, Ichiba S. A Case of Leptospirosis-Associated Severe Pulmonary Hemorrhagic Syndrome Successfully Treated with Venovenous Extracorporeal Membrane Oxygenation. Case Rep Crit Care. 2017;2017:5369267. doi: 10.1155/2017/5369267. Epub 2017 Oct 25. PMID 29312788
- [Background] Cantwell T, Ferre A, Van Sint Jan N, Blamey R, Dreyse J, Baeza C, Diaz R, Regueira T. Leptospirosis-associated catastrophic respiratory failure supported by extracorporeal membrane oxygenation. J Artif Organs. 2017 Dec;20(4):371-376. doi: 10.1007/s10047-017-0998-x. Epub 2017 Oct 10. PMID 29019017
- [Background] Vandroux D, Chanareille P, Delmas B, Gauzere BA, Allou N, Raffray L, Jaffar-Bandjee MC, Martinet O, Ferdynus C, Jabot J. Acute respiratory distress syndrome in leptospirosis. J Crit Care. 2019 Jun;51:165-169. doi: 10.1016/j.jcrc.2019.02.018. Epub 2019 Feb 18. PMID 30831550
- [Background] Saadah NH, van der Bom JG, Wiersum-Osselton JC, Richardson C, Middelburg RA, Politis C, Renaudier P, Robillard P, Schipperus MR. Comparing transfusion reaction risks for various plasma products - an analysis of 7 years of ISTARE haemovigilance data. Br J Haematol. 2018 Mar;180(5):727-734. doi: 10.1111/bjh.15082. Epub 2018 Jan 9. PMID 29318576
- [Background] Kracalik I, Mowla S, Basavaraju SV, Sapiano MRP. Transfusion-related adverse reactions: Data from the National Healthcare Safety Network Hemovigilance Module - United States, 2013-2018. Transfusion. 2021 May;61(5):1424-1434. doi: 10.1111/trf.16362. Epub 2021 Apr 20. PMID 33880771
- [Background] van den Akker TA, Grimes ZM, Friedman MT. Transfusion-Associated Circulatory Overload and Transfusion-Related Acute Lung Injury. Am J Clin Pathol. 2021 Sep 8;156(4):529-539. doi: 10.1093/ajcp/aqaa279. PMID 33822854
- [Background] Pandey S, Vyas GN. Adverse effects of plasma transfusion. Transfusion. 2012 May;52 Suppl 1(Suppl 1):65S-79S. doi: 10.1111/j.1537-2995.2012.03663.x. PMID 22578374
- [Background] Carman M, Uhlenbrock JS, McClintock SM. CE: A Review of Current Practice in Transfusion Therapy. Am J Nurs. 2018 May;118(5):36-44. doi: 10.1097/01.NAJ.0000532808.81713.fc. PMID 29664740
- [Background] Combes A, Peek GJ, Hajage D, Hardy P, Abrams D, Schmidt M, Dechartres A, Elbourne D. ECMO for severe ARDS: systematic review and individual patient data meta-analysis. Intensive Care Med. 2020 Nov;46(11):2048-2057. doi: 10.1007/s00134-020-06248-3. Epub 2020 Oct 6. PMID 33021684
- [Background] Fonseka CL, Lekamwasam S. Role of Plasmapheresis and Extracorporeal Membrane Oxygenation in the Treatment of Leptospirosis Complicated with Pulmonary Hemorrhages. J Trop Med. 2018 Dec 2;2018:4520185. doi: 10.1155/2018/4520185. eCollection 2018. PMID 30631369
- [Background] Heymann M, Schorer R, Putzu A. Mortality and adverse events of hemoadsorption with CytoSorb(R) in critically ill patients: A systematic review and meta-analysis of randomized controlled trials. Acta Anaesthesiol Scand. 2022 Oct;66(9):1037-1050. doi: 10.1111/aas.14115. Epub 2022 Jul 18. PMID 35788557
- [Background] Li X, Liu C, Mao Z, Qi S, Song R, Zhou F. Effectiveness of polymyxin B-immobilized hemoperfusion against sepsis and septic shock: A systematic review and meta-analysis. J Crit Care. 2021 Jun;63:187-195. doi: 10.1016/j.jcrc.2020.09.007. Epub 2020 Sep 18. PMID 33012579
- [Background] Ronco C, Bellomo R. Hemoperfusion: technical aspects and state of the art. Crit Care. 2022 May 12;26(1):135. doi: 10.1186/s13054-022-04009-w. PMID 35549999
- [Background] Landini S, Coli U, Lucatello S, Bazzato G. Plasma exchange in severe leptospirosis. Lancet. 1981 Nov 14;2(8255):1119-20. doi: 10.1016/s0140-6736(81)91329-5. No abstract available. PMID 6118571
- [Background] Chen YS, Cheng SL, Wang HC, Yang PC. Successful treatment of pulmonary hemorrhage associated with leptospirosis and scrub typhus coinfection by early plasma exchange. J Formos Med Assoc. 2007 Feb;106(2 Suppl):S1-6. doi: 10.1016/s0929-6646(09)60344-2. PMID 17493889
- [Background] Bourquin V, Ponte B, Hirschel B, Pugin J, Martin PY, Saudan P. Severe leptospirosis with multiple organ failure successfully treated by plasma exchange and high-volume hemofiltration. Case Rep Nephrol. 2011;2011:817414. doi: 10.1155/2011/817414. Epub 2011 Sep 13. PMID 24527237
- [Background] Cerdas-Quesada C. Potential benefits of plasma exchange by apheresis on the treatment of severe Icteric Leptospirosis: case report and literature review. Transfus Apher Sci. 2011 Oct;45(2):191-4. doi: 10.1016/j.transci.2011.07.012. Epub 2011 Sep 1. PMID 21889407
- [Background] Taylor D, Karamadoukis L. Plasma exchange in severe leptospirosis with multi-organ failure: a case report. J Med Case Rep. 2013 Jun 28;7:169. doi: 10.1186/1752-1947-7-169. PMID 23809518
- [Background] Ekinci F, Yildizdas RD, Horoz OO, Alabaz D, Tolunay I, Petmezci E. Treatment of severe leptospirosis with therapeutic plasma exchange in a pediatric patient. Turk J Pediatr. 2018;60(5):566-570. doi: 10.24953/turkjped.2018.05.015. PMID 30968640
- [Background] Huang Z, Wang SR, Yang ZL, Liu JY. Effect on extrapulmonary sepsis-induced acute lung injury by hemoperfusion with neutral microporous resin column. Ther Apher Dial. 2013 Aug;17(4):454-61. doi: 10.1111/j.1744-9987.2012.01083.x. Epub 2012 Jun 21. PMID 23931889
- [Background] Butylin VYu, Chepkij LP, Lenartovich LS. Urgent hemosorption in leptospirosis. Biomater Artif Cells Artif Organs. 1987;15(1):249-56. doi: 10.3109/10731198709118525. PMID 3449141
- [Background] Putzu A, Schorer R, Lopez-Delgado JC, Cassina T, Landoni G. Blood Purification and Mortality in Sepsis and Septic Shock: A Systematic Review and Meta-analysis of Randomized Trials. Anesthesiology. 2019 Sep;131(3):580-593. doi: 10.1097/ALN.0000000000002820. PMID 31246600
- [Background] Girardot T, Schneider A, Rimmele T. Blood Purification Techniques for Sepsis and Septic AKI. Semin Nephrol. 2019 Sep;39(5):505-514. doi: 10.1016/j.semnephrol.2019.06.010. PMID 31514914
- [Background] Castiblanco-Valencia MM, Fraga TR, Silva LB, Monaris D, Abreu PA, Strobel S, Jozsi M, Isaac L, Barbosa AS. Leptospiral immunoglobulin-like proteins interact with human complement regulators factor H, FHL-1, FHR-1, and C4BP. J Infect Dis. 2012 Mar 15;205(6):995-1004. doi: 10.1093/infdis/jir875. Epub 2012 Jan 30. PMID 22291192
- [Background] Muthuppalaniappan VM, Rajakariar R, Blunden MJ. Leptospirosis presenting as haemolytic uraemic syndrome: a case report. BMC Nephrol. 2018 Jan 29;19(1):20. doi: 10.1186/s12882-018-0817-5. PMID 29378539
- [Background] Fraga TR, Barbosa AS, Isaac L. Leptospirosis: aspects of innate immunity, immunopathogenesis and immune evasion from the complement system. Scand J Immunol. 2011 May;73(5):408-19. doi: 10.1111/j.1365-3083.2010.02505.x. PMID 21204903
- [Background] Cinco M. New insights into the pathogenicity of leptospires: evasion of host defences. New Microbiol. 2010 Oct;33(4):283-92. PMID 21213586
- [Background] Fremeaux-Bacchi V, Dragon-Durey MA, Blouin J, Vigneau C, Kuypers D, Boudailliez B, Loirat C, Rondeau E, Fridman WH. Complement factor I: a susceptibility gene for atypical haemolytic uraemic syndrome. J Med Genet. 2004 Jun;41(6):e84. doi: 10.1136/jmg.2004.019083. No abstract available. PMID 15173250
- [Background] Crovetto F, Borsa N, Acaia B, Nishimura C, Frees K, Smith RJ, Peyvandi F, Palla R, Cugno M, Tedeschi S, Castorina P, Somigliana E, Ardissino G, Fedele L. The genetics of the alternative pathway of complement in the pathogenesis of HELLP syndrome. J Matern Fetal Neonatal Med. 2012 Nov;25(11):2322-5. doi: 10.3109/14767058.2012.694923. Epub 2012 Jun 7. PMID 22594569
- [Background] Tsiftsoglou SA, Willis AC, Li P, Chen X, Mitchell DA, Rao Z, Sim RB. The catalytically active serine protease domain of human complement factor I. Biochemistry. 2005 Apr 26;44(16):6239-49. doi: 10.1021/bi047680t. PMID 15835912
- [Background] Goswami RP, Goswami RP, Basu A, Tripathi SK, Chakrabarti S, Chattopadhyay I. Predictors of mortality in leptospirosis: an observational study from two hospitals in Kolkata, eastern India. Trans R Soc Trop Med Hyg. 2014 Dec;108(12):791-6. doi: 10.1093/trstmh/tru144. Epub 2014 Oct 30. PMID 25359320
- [Background] Abgueguen P, Delbos V, Blanvillain J, Chennebault JM, Cottin J, Fanello S, Pichard E. Clinical aspects and prognostic factors of leptospirosis in adults. Retrospective study in France. J Infect. 2008 Sep;57(3):171-8. doi: 10.1016/j.jinf.2008.06.010. Epub 2008 Jul 24. PMID 18656263
- [Background] Lee N, Kitashoji E, Koizumi N, Lacuesta TLV, Ribo MR, Dimaano EM, Saito N, Suzuki M, Ariyoshi K, Parry CM. Building prognostic models for adverse outcomes in a prospective cohort of hospitalised patients with acute leptospirosis infection in the Philippines. Trans R Soc Trop Med Hyg. 2017 Dec 1;111(12):531-539. doi: 10.1093/trstmh/try015. PMID 29518223
- [Background] Wang HK, Lee MH, Chen YC, Hsueh PR, Chang SC. Factors associated with severity and mortality in patients with confirmed leptospirosis at a regional hospital in northern Taiwan. J Microbiol Immunol Infect. 2020 Apr;53(2):307-314. doi: 10.1016/j.jmii.2018.05.005. Epub 2018 Jun 6. PMID 29934034
- [Background] Smith S, Kennedy BJ, Dermedgoglou A, Poulgrain SS, Paavola MP, Minto TL, Luc M, Liu YH, Hanson J. A simple score to predict severe leptospirosis. PLoS Negl Trop Dis. 2019 Feb 13;13(2):e0007205. doi: 10.1371/journal.pntd.0007205. eCollection 2019 Feb. PMID 30759081
- [Background] Marotto PC, Ko AI, Murta-Nascimento C, Seguro AC, Prado RR, Barbosa MC, Cleto SA, Eluf-Neto J. Early identification of leptospirosis-associated pulmonary hemorrhage syndrome by use of a validated prediction model. J Infect. 2010 Mar;60(3):218-23. doi: 10.1016/j.jinf.2009.12.005. Epub 2009 Dec 21. PMID 20026189
- [Background] Vieira SR, Brauner JS. Leptospirosis as a cause of acute respiratory failure: clinical features and outcome in 35 critical care patients. Braz J Infect Dis. 2002 Jun;6(3):135-9. doi: 10.1590/s1413-86702002000300006. Epub 2003 Mar 6. PMID 12144750
- [Background] Marotto PC, Nascimento CM, Eluf-Neto J, Marotto MS, Andrade L, Sztajnbok J, Seguro AC. Acute lung injury in leptospirosis: clinical and laboratory features, outcome, and factors associated with mortality. Clin Infect Dis. 1999 Dec;29(6):1561-3. doi: 10.1086/313501. PMID 10585813
- [Background] Herath N, Uluwattage W, Weliwitiya T, Karunanayake L, Lekamwasam S, Ratnatunga N, Karunanayake P, Wickramasinghe S, Patabendi S, Senaviratne S, Agampodi S. Sequel and therapeutic modalities of leptospirosis associated severe pulmonary haemorrhagic syndrome (SPHS); a Sri Lankan experience. BMC Infect Dis. 2019 May 22;19(1):451. doi: 10.1186/s12879-019-4094-0. PMID 31113404
- [Background] Gulati S, Gulati A. Pulmonary manifestations of leptospirosis. Lung India. 2012 Oct;29(4):347-53. doi: 10.4103/0970-2113.102822. PMID 23243349
- [Background] Gouveia EL, Metcalfe J, de Carvalho AL, Aires TS, Villasboas-Bisneto JC, Queirroz A, Santos AC, Salgado K, Reis MG, Ko AI. Leptospirosis-associated severe pulmonary hemorrhagic syndrome, Salvador, Brazil. Emerg Infect Dis. 2008 Mar;14(3):505-8. doi: 10.3201/eid1403.071064. PMID 18325275
- [Background] World Health Organization (WHO). (2003). Human leptospirosis: guidance for diagnosis, surveillance, and control. World Health Organization, Geneva, Switzerland.
- [Background] Sollberger G, Choidas A, Burn GL, Habenberger P, Di Lucrezia R, Kordes S, Menninger S, Eickhoff J, Nussbaumer P, Klebl B, Kruger R, Herzig A, Zychlinsky A. Gasdermin D plays a vital role in the generation of neutrophil extracellular traps. Sci Immunol. 2018 Aug 24;3(26):eaar6689. doi: 10.1126/sciimmunol.aar6689. PMID 30143555
- [Background] Scharrig E, Carestia A, Ferrer MF, Cedola M, Pretre G, Drut R, Picardeau M, Schattner M, Gomez RM. Neutrophil Extracellular Traps are Involved in the Innate Immune Response to Infection with Leptospira. PLoS Negl Trop Dis. 2015 Jul 10;9(7):e0003927. doi: 10.1371/journal.pntd.0003927. eCollection 2015. PMID 26161745
- [Background] Cagliero J, Villanueva SYAM, Matsui M. Leptospirosis Pathophysiology: Into the Storm of Cytokines. Front Cell Infect Microbiol. 2018 Jun 20;8:204. doi: 10.3389/fcimb.2018.00204. eCollection 2018. PMID 29974037
- [Background] Trivedi SV, Vasava AH, Bhatia LC, Patel TC, Patel NK, Patel NT. Plasma exchange with immunosuppression in pulmonary alveolar haemorrhage due to leptospirosis. Indian J Med Res. 2010 Mar;131:429-33. PMID 20418558
- [Background] Segura ER, Ganoza CA, Campos K, Ricaldi JN, Torres S, Silva H, Cespedes MJ, Matthias MA, Swancutt MA, Lopez Linan R, Gotuzzo E, Guerra H, Gilman RH, Vinetz JM; Peru-United States Leptospirosis Consortium. Clinical spectrum of pulmonary involvement in leptospirosis in a region of endemicity, with quantification of leptospiral burden. Clin Infect Dis. 2005 Feb 1;40(3):343-51. doi: 10.1086/427110. Epub 2005 Jan 10. PMID 15668855
- [Background] Haake DA, Levett PN. Leptospirosis in humans. Curr Top Microbiol Immunol. 2015;387:65-97. doi: 10.1007/978-3-662-45059-8_5. PMID 25388133
- [Background] Bharti AR, Nally JE, Ricaldi JN, Matthias MA, Diaz MM, Lovett MA, Levett PN, Gilman RH, Willig MR, Gotuzzo E, Vinetz JM; Peru-United States Leptospirosis Consortium. Leptospirosis: a zoonotic disease of global importance. Lancet Infect Dis. 2003 Dec;3(12):757-71. doi: 10.1016/s1473-3099(03)00830-2. PMID 14652202
- [Background] Costa F, Hagan JE, Calcagno J, Kane M, Torgerson P, Martinez-Silveira MS, Stein C, Abela-Ridder B, Ko AI. Global Morbidity and Mortality of Leptospirosis: A Systematic Review. PLoS Negl Trop Dis. 2015 Sep 17;9(9):e0003898. doi: 10.1371/journal.pntd.0003898. eCollection 2015. PMID 26379143
- [Background] Chavez JR, Danguilan RA, Arakama MI, Garcia JKG, So R, Chua E. A case of leptospirosis with acute respiratory failure and acute kidney injury treated with simultaneous extracorporeal membrane oxygenation and haemoperfusion. BMJ Case Rep. 2019 May 29;12(5):e229582. doi: 10.1136/bcr-2019-229582. PMID 31147412

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT07127718/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT07127718/ICF_001.pdf